CLINICAL TRIAL: NCT04194203
Title: A Phase III, Randomized, Double-Blind Study of Bevacizumab, Carboplatin, and Paclitaxel or Pemetrexed With or Without Atezolizumab in Chemotherapy-Naïve Patients With Stage IV Non-Squamous Non-Small Cell Lung Cancer (IMpower151)
Brief Title: A Study of Bevacizumab, Carboplatin, and Paclitaxel or Pemetrexed With or Without Atezolizumab in Chemotherapy-Naïve Patients With Stage IV Non-Squamous Non-Small Cell Lung Cancer (IMpower151)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO30157
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Bevacizumab; Paclitaxel; Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive atezolizumab, bevacizumab, paclitaxel or pemetrexed, and carboplatin (in this order) by intravenous (IV) injection on Day 1 of each 21-day cycle for 4 cycles in the induction treatment. In the maintenance phase, participants will be treated with atezolizumab, bevacizumab and pemetrexed (if given in the induction phase) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Carboplatin
- Treatment B (Placebo Comparator): Participants will receive placebo, bevacizumab, paclitaxel or pemetrexed, and carboplatin (in this order) by intravenous (IV) injection on Day 1 of each 21-day cycle for 4 cycles in the induction treatment. In the maintenance phase, participants will be treated with placebo, bevacizumab and pemetrexed (if given in the induction phase) until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Placebo; Drug: Bevacizumab; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.
  Other Names: Tecentriq
  Arms: Treatment A
Drug: Placebo — Placebo matching to atezolizumab will be administered by IV infusion at a fixed dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.
  Arms: Treatment B
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a dose of 15 mg/kg on Day 1 of each 21-day cycle.
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel will be administered by IV infusion at a dose of 175 mg/m2.
Drug: Pemetrexed — Pemetrexed will be administered by IV infusion at a dose of 500 mg/m2.
Drug: Carboplatin — Carboplatin will be administered by IV infusion to achieve an initial target AUC of 6 mg/mL/min.

SUMMARY:
This study will evaluate the efficacy and safety of atezolizumab when given in combination with bevacizumab, investigator's choice of either paclitaxel or pemetrexed, and carboplatin compared with placebo given in combination with bevacizumab, paclitaxel or pemetrexed, and carboplatin in patients with chemotherapy-naive, Stage IV non-squamous Non-Small Cell Lung Cancer (NSCLC). The study will be conducted in two phases: Induction Phase and Maintenance Phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IV non-squamous NSCLC
* No prior treatment for Stage IV non-squamous NSCLC, with the following exceptions: (1) Patients with a sensitizing mutation in the EGFR gene must have experienced disease progression (during or after treatment) or were intolerant to treatment with one or more EGFR TKIs, such as erlotinib, gefitinib, afatinib, dacomitinib, and osimertinib, or another EGFR TKI appropriate for the treatment of EGFR-mutant NSCLC. Patients who have progressed on or were intolerant to first-line osimertinib or other third-generation EGFR TKIs are eligible. Patients who have progressed on or were intolerant to first- or second-generation EGFR TKIs, such as erlotinib, gefitinib, afatinib, dacomitinib, and who have no evidence of the EGFR T790M mutation in the tumor tissue after TKI therapy are eligible. Patients who have progressed on or were intolerant to first- or second-generation EGFR TKIs and who have evidence of the T790M mutation in their tumor tissue must have also progressed on or were intolerant to osimertinib to be eligible. (2) Patients with an ALK gene rearrangement must have experienced disease progression or were intolerant to treatment with one or more ALK inhibitors, such as crizotinib, alectinib, ceritinib, brigatinib, ensartinib and lorlatinib that are appropriate for the treatment of NSCLC that has an ALK gene rearrangement.
* Availability of a representative tumor specimen that is suitable for the determination of PD-L1 status, as well as the presence of EGFR mutations and ALK gene rearrangements, via central testing.
* Treatment-free interval of at least 6 months from randomization since the last chemotherapy, radiotherapy, or chemoradiotherapy treatment for patients who have received prior neoadjuvant and/or adjuvant chemotherapy, radiotherapy, or chemoradiotherapy with curative intent for non-metastatic disease
* Measurable disease, as defined by RECIST v1.1
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Life expectancy >=3 months
* Adequate hematologic and end-organ function
* Negative HIV test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
* History of malignancy other than NSCLC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Prior allogeneic stem cell or solid organ transplantation
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with any approved anti-cancer therapy or investigational therapy within 28 days prior to initiation of study treatment, except for treatment with TKI that should be discontinued for at least 8 days or for approximately 5 x half-life, whichever is the longer, before the first dose of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab or 6 months after the final dose of bevacizumab, carboplatin, pemetrexed, and paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in the intent to treat (ITT) population, as determined by the investigator | Randomization until the first occurence of disease progression or death from any cause, whichever occures first (up to approximately 33 months)
  PFS after randomization, defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Overall Survival (OS) in the ITT population | Randomization to death from any cause (up to approximately 33 months)
  OS after randomization, defined as the time from randomization to death from any cause.
PFS in the ITT population, as determined by IRF | Randomization until the first occurence of disease progression or death from any cause, whichever occures first (up to approximately 33 months)
  PFS after randomizationdefined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the an Independent Review Facility (IRF) according to RECIST v1.1
PFS in subgroup of participants with PD-L1 Expression, as determined by the investigator | Randomization until the first occurence of disease progression or death from any cause, whichever occures first (up to approximately 33 months)
  PFS after randomization as determined by the investigator according to RECIST v1.1 in the subgroup of patients with PD-L1 expression defined by the SP263 immunohistochemistry (IHC) assay.
PFS in the subgroup of participants with genomic alterations in EGFR or ALK gene, as determined by the investigator | Randomization until the first occurence of disease progression or death from any cause, whichever occures first (up to approximately 33 months)
  PFS after randomization as determined by the investigator according to RECIST v1.1 in the subgroup of patients with genomic alterations in EGFR (i.e., sensitizing EGFR mutations) or ALK gene.
Objective Response Rate (ORR) in the ITT population | Randomization until disease progression or death, which ever occurs first (up to approximately 33 months)
  ORR, defined as the proportion of patients with a complete response (CR) or partial response (PR) on two consecutive occasions >=4 weeks apart, as determined by the investigator according to RECIST v1.1.
Duration of response (DOR) in the ITT population | Randomization until the first occurence of a documented objective response to disease progression or death from any cause, whichever occures first (up to approximately 33 months)
  DOR defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Time to Confirmed Deterioration (TTCD) in physical functioning in the ITT population | Randomization up until approximately 33 months
  (TTCD) in physical functioning, defined as the time from randomization to the first observed >=10-point decrease in the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) for cancer linearly transformed physical functioning scale score that is sustained for two consecutive assessments or an initial clinically meaningful decrease above baseline followed by death within three weeks.
Percentage of Participants With Adverse Events | Randomization up to approximately 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- China (23):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital; Oncology Department, Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - The 900th Hospital of PLA joint service support force, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Nan Tong Tumor Hospital, Nantong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Liaoning cancer Hospital & Institute, Shenyang
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center; Cancer Center, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).